CLINICAL TRIAL: NCT02380612
Title: Demonstration of the Safety and Effectiveness of ReCell® Combined With Meshed Skin Graft for Reduction of Donor Area in the Treatment of Acute Burn Injuries
Brief Title: ReCell® Combined With Meshed Skin Graft in the Treatment of Acute Burn Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avita Medical (Industry)
Collaborators: MedDRA Assistance Inc (Unknown); Advanced Clinical Research Services, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTP001-6
Record Dates: First submitted 2015-02-17; First posted 2015-03-05 (Estimated); Results first posted 2021-02-23 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Burns
Keywords: Second Degree Burn Injuries
MeSH Terms: conditions — Burns | interventions — Skin Transplantation

STUDY DESIGN:
Masking Description: The participant and blinded evaluator will be not be told which treatment area received which treatment (RECELL or Control).
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Participants (within patient control) (Experimental): All subjects will receive both ReCell and skin graft. Each patient serves as their own control. Their study treatment area (burn injury) will be divided into Area A and Area B. Investigational treatment will be randomly allocated to either Area A or Area B
  Interventions: Device: ReCell Treatment; Procedure: Skin Graft

INTERVENTIONS:
Device: ReCell Treatment
Procedure: Skin Graft

SUMMARY:
This is a randomized, within-subject controlled study to compare the clinical performance of the ReCell device when used as an adjunct to meshed skin graft in subjects requiring skin grafts for closure of burn injuries. Co-primary effectiveness endpoints include: (1) confirmed treatment area closure (i.e., healing) prior to or at 8 weeks as assessed by a blinded evaluator, and (2) a comparison of the actual expansion ratio, computed as the ratio of measured treated area to the measured donor site area, achieved for the ReCell-treated and control treatment areas. Safety will be evaluated in terms of long-term durability, scar outcomes and treatment-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. The subject requires skin grafting as a result of an acute thermal burn injury (i.e. injuries caused by exposure of the skin to fire/flames, excessive heat, hot steam or water).
2. The area of total burn injury is 5-50% TBSA inclusive.
3. Two areas requiring skin grafting, each at least 300cm2 (or 600cm2 contiguous), excluding hand/face and joints.
4. The subject is at least 5 years of age.
5. The subject (or family, for those under 18 years of age) is willing and able to complete all followup evaluations required by the study protocol.
6. The subject is to abstain from any other treatment of the wound(s) for the duration of the study unless medically necessary.
7. The subject agrees to abstain from enrollment in any other interventional clinical trial for the duration of the study.
8. The subject and/or guardian are able to read and understand instructions and give informed, voluntary, written consent.

Exclusion Criteria:

1. The subject's burn injuries were caused by chemicals, electricity, and/or radioactive substances.
2. The subject is unable to follow the protocol.
3. The subject has other concurrent conditions that in the opinion of the investigator may compromise patient safety or study objectives.
4. The subject has a known hypersensitivity to trypsin or compound sodium lactate for irrigation (Hartmann's) solution.
5. Life expectancy is less than 1 year.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01-26 (Actual); Primary Completion 2016-01-21 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James H Holmes, IV, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (7):
- United States (7):
  - Arizona Burn Center at Maricopa Medical Center, Phoenix, Arizona
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Tampa General Hospital, Tampa, Florida
  - North Carolina Jaycee Burn Center, Chapel Hill, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - USAISR - US Army Institute of Surgical Research, Fort Sam Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: All Participants (Within Patient Control): Every subject received both interventions (RECELL and CONTROL) such that each subject served as their own control. Each subject's study treatment area (burn injury) was divided into Area A and Area B before thee areas (A and B) were randomly assigned to receive CONTROL (grafting consistent with the pre-identified graft plan) or RECELL (RECELL-generated cell suspension applied over a graft more widely meshed than identified in the pre-specified graft plan).
Period: Overall Study
Arm/Group | Experimental: All Participants (Within Patient Control)
Started | 30
Completed | 27
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Experimental: All Participants (Within Patient Control): All subjects receive both ReCell treatment and autograft (Area A and Area B). Each subject serves as their own control. Wound regions were randomly assigned to receive an autograft consistent with the investigator's pre-identified graft plan (Control) or to receive application of the ReCell-generated cell suspension over an autograft more widely meshed than identified in the investigator's pre-specified graft plan (ReCell-treated).
Arm/Group | Experimental: All Participants (Within Patient Control)
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 25
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (15.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 20
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Confirmed Treatment Area Closure of RECELL-treated Wounds Compared to Control (Non-inferiority)
Description: Complete wound closure is defined as skin re-epithelialization without drainage, confirmed at two consecutive study visits at least 2 weeks apart by direct visualization by a qualified clinician blinded to treatment assignment. The incidence of complete wound closure is hypothesized to be non-inferior for RECELL-treated areas as compared to control areas.
Time Frame: Prior to or at 8 weeks
Population: Per Protocol Population
Measure: Count of Participants; unit: Participants
Groups:
- RECELL-Treated: Wound received application of the RECELL-generated cell suspension over an autograft more widely meshed than identified in the investigator's pre-specified graft plan (RECELL-treated).
- Control: Wound received an autograft consistent with the investigator's pre-identified graft plan (Control).
Arm/Group | RECELL-Treated | Control
Number analyzed (Participants) | 26 | 26
Participants
  Confirmed Closure | 24 | 22
  Not Healed | 2 | 4

2. Primary Outcome: Actual Expansion Ratios (Treatment Area to Donor Site Area, Inclusive of Donor Skin Needed for Secondary Treatments)
Description: For this second co-primary endpoint, it is hypothesized that the expansion ratio associated with the RECELL treatment area will be superior to that of the control, i.e. less donor skin will be required for RECELL-treated areas compared with the control areas.
Time Frame: Prior to or at 8 weeks
Population: Intent-to-Treat Population (primary analysis)
Measure: Geometric Mean (Standard Deviation); unit: cm2
Arm/Group | RECELL-Treated | Control
Number analyzed (Participants) | 30 | 30
cm2 | 1.9657 (2.0415) | 1.3486 (1.4143)
Statistical Analysis 1: Comparison: RECELL-Treated vs Control; Test type: Other; Geometric Mean Ratio = 1.4575

3. Secondary Outcome: Observer Overall Patient and Observer Scar Assessment Scale ( POSAS) Opinion Score
Description: The observer component of the Patient and Observer Scar Assessment Scale (POSAS) questionnaire required the blinded evaluator to provide an overall opinion of the treatment area compared to normal skin, scored from 1 (normal skin) to 10 (worst imaginable scar).
Time Frame: At 24 Week
Population: Per-Protocol Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RECELL-Treated | Control
Number analyzed (Participants) | 26 | 26
units on a scale | 2.6 (1.20) | 2.5 (1.42)

4. Secondary Outcome: Patient's Satisfaction/Treatment Preference
Time Frame: At 24 Week
Population: Per-Protocol Population
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects: Every subject received both interventions (RECELL and CONTROL)
Arm/Group | All Subjects
Number analyzed (Participants) | 26
Participants
  Preferred RECELL | 12
  Preferred CONTROL | 12
  No Preference | 2

5. Secondary Outcome: Patient Overall Patient and Observer Scar Assessment Scale (POSAS) Opinion Score
Description: The patient component of the Patient Overall Patient and Observer Scar Assessment Scale (POSAS) questionnaire required the patient to provide an overall opinion of the treatment area compared to normal skin, scored from 1 (normal skin) to 10 (worst imaginable scar). T
Time Frame: Week 24
Population: Per-Protocol Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RECELL-Treated | CONTROL
Number analyzed (Participants) | 25 | 25
units on a scale | 5.2 (2.76) | 5.1 (2.96)

ADVERSE EVENTS:
Time Frame: 52 Weeks
Arm/Group | Experimental: All Participants (Within Patient Control)
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 12/30
Other Adverse Events (participants affected / at risk) | 26/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: All Participants (Within Patient Control) (N=30)
Failed Skin Graft (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Graft Loss (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Re-grafting Due to Graft Failure (Injury, poisoning and procedural complications) | 1 (1) — CONTROL
Surgery for Failed Skin Graft (Injury, poisoning and procedural complications) | 1 (1) — CONTROL
Graft Loss to Left Lower Extremity (LLE) (Injury, poisoning and procedural complications) | 1 (1) — CONTROL
Re-Grafting Due to Graft Failure (Injury, poisoning and procedural complications) | 1 (1) — NON-STUDY AREA
Severe Contracture left hand, left wrist, left fingers and left lower eyelid (Musculoskeletal and connective tissue disorders) | 1 (1) — NON-STUDY AREA
Open Wound Left Elbow (Injury, poisoning and procedural complications) | 1 (1) — NON-STUDY AREA
Increased Elbow Pain, Right (Musculoskeletal and connective tissue disorders) | 1 (1) — NON-STUDY AREA
Inability to Move Right Elbow (Musculoskeletal and connective tissue disorders) | 1 (1) — NON-STUDY AREA
Intractable Pain Right Arm (Musculoskeletal and connective tissue disorders) | 1 (1) — NON-STUDY AREA
Cellulitis Left Index Finger (Infections and infestations) | 1 (1) — NON-STUDY AREA
Cellulitis to Non-Study Donor Site (Infections and infestations) | 1 (1) — NON-STUDY AREA
Graft Loss (Injury, poisoning and procedural complications) | 1 (1) — NON-STUDY AREA
Graft Shearing/Loss to Left Calf (Injury, poisoning and procedural complications) | 1 (1) — NON-STUDY AREA
Patient Concern for Infection (General disorders) | 1 (1) — NON-STUDY AREA
Nausea (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1)
Acute respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Right Frontotemporal Subarachnoid Hemorrhage (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: All Participants (Within Patient Control) (N=30)
Itching (Skin and subcutaneous tissue disorders) | 6 (6) — RECELL
Pain/Soreness Under Right Arm (Musculoskeletal and connective tissue disorders) | 1 (1) — RECELL
Chronic Pain (General disorders) | 1 (1) — RECELL
Scar Revision (Surgical and medical procedures) | 1 (1) — RECELL
Neuropathic Pain (Nervous system disorders) | 1 (1) — RECELL
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) — RECELL
Burning (Nervous system disorders) | 1 (1) — RECELL
Shearing of Graft on Site A 0.9x1 cm (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Delayed Healing (General disorders) | 1 (1) — RECELL
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) — RECELL
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — RECELL
Increased Pain (General disorders) | 1 (1) — RECELL
Abrasion (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Scratch on Back (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Small area of graft loss on anterior right lower extremity (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Chronic non-healing wounds to RLE secondary to DM type 1 (Skin and subcutaneous tissue disorders) | 1 (1) — RECELL
Graft Loss Posterior Back (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Itching (Skin and subcutaneous tissue disorders) | 6 (6) — CONTROL
Mildly Infected (Infections and infestations) | 1 (1) — CONTROL
Chronic Pain (General disorders) | 1 (1) — CONTROL
Scar Revision (Surgical and medical procedures) | 1 (1) — CONTROL
Neuropathic Pain (Nervous system disorders) | 1 (1) — CONTROL
Graft Loss (Injury, poisoning and procedural complications) | 1 (1) — CONTROL
Delayed Healing (General disorders) | 3 (3) — CONTROL
Ossification (Musculoskeletal and connective tissue disorders) | 1 (1) — CONTROL
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) — CONTROL
Burning (Nervous system disorders) | 1 (1) — CONTROL
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) — CONTROL
Abrasion to shin (Injury, poisoning and procedural complications) | 1 (1) — CONTROL
White creamy exudates left lower leg (General disorders) | 1 (1) — CONTROL
Infection of the L Lower Leg (Infections and infestations) | 1 (2) — CONTROL
Chronic non-healing wounds to LLE secondary to DM type 1 (Skin and subcutaneous tissue disorders) | 1 (1) — CONTROL
Graft loss posterior back (Injury, poisoning and procedural complications) | 1 (1) — CONTROL
Itching (Skin and subcutaneous tissue disorders) | 2 (2) — DONOR SITE
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) — DONOR SITE
Blisters (Skin and subcutaneous tissue disorders) | 1 (1) — DONOR SITE
Left thigh donor site with purulent drainage and open areas (Infections and infestations) | 1 (1) — DONOR SITE
Pain right hand (Musculoskeletal and connective tissue disorders) | 1 (1) — NON-STUDY AREA
Itching (Skin and subcutaneous tissue disorders) | 4 (4) — NON-STUDY AREA
Chronic pain (General disorders) | 1 (1) — NON-STUDY AREA
Scar revision (Surgical and medical procedures) | 1 (1) — NON-STUDY AREA
Neuropathic pain (Nervous system disorders) | 1 (1) — NON-STUDY AREA
Heterotrophic ossification (Musculoskeletal and connective tissue disorders) | 1 (1) — NON-STUDY AREA
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) — NON-STUDY AREA
Burning (Nervous system disorders) | 1 (1) — NON-STUDY AREA
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) — NON-STUDY AREA
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — NON-STUDY AREA
Contracture, right hand (Musculoskeletal and connective tissue disorders) | 1 (1) — NON-STUDY AREA
Blisters to left thigh non-study donor (Skin and subcutaneous tissue disorders) | 1 (1) — NON-STUDY AREA
Blisters to right thigh non-study graft (Skin and subcutaneous tissue disorders) | 1 (1) — NON-STUDY AREA
Non-healing wound to posterior left upper arm (General disorders) | 1 (1) — NON-STUDY AREA
Abrasion to knee (Injury, poisoning and procedural complications) | 1 (1) — NON-STUDY AREA
Scratch at the back (Injury, poisoning and procedural complications) | 1 (1) — NON-STUDY AREA
Contact dermatitis at neck and upper back (Skin and subcutaneous tissue disorders) | 1 (1) — NON-STUDY AREA
Graft loss l breast (Injury, poisoning and procedural complications) | 1 (1) — NON-STUDY AREA
Medial left upper arm graft loss (Injury, poisoning and procedural complications) | 1 (1) — NON-STUDY AREA
Arm burn cellulitis (Infections and infestations) | 1 (1) — NON-STUDY AREA
Graft loss chest wall at inner axilla (Injury, poisoning and procedural complications) | 1 (1) — NON-STUDY AREA
Confusion (Psychiatric disorders) | 1 (1)
Klebsiella Pneumonia (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No